CLINICAL TRIAL: NCT05710133
Title: The Food-effect of a Standardized Dutch Breakfast on the Pharmacokinetics of Oral Alectinib (Alecensa®) Using a Stable Isotopically Labelled Microtracer Approach
Brief Title: The Food-effect on Alectinib Pharmacokinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N20FEA; 2021-006957-69 (EudraCT Number)
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: NSCLC
MeSH Terms: interventions — Food

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- alectinib-d6 (Other): Patients will receive one single dose of alectinib-d6 (100 µg) orally on day 1 and 9.
  Interventions: Other: food; Other: fast

INTERVENTIONS:
Other: food — alectinib-d6 will be administered with breakfast on day 1 to determine the food-effect
  Other Names: food state
Other: fast — alectinib-d6 will be administered after an overnight fast of minimal 10 hours on day 9 to determine the food-effect
  Other Names: fast state

SUMMARY:
The goal of this food-effect study on Alectinib pharmacokinetics is to learn about the food effect of alectinib. The main question aims to answer is:

• To determine the food-effect of a standardized Dutch breakfast on the pharmacokinetics of oral alectinib (Alecensa®), especially Peak Plasma Concentration (Cmax), Area under the plasma concentration versus time curve (AUC) and relative bioavailability, at steady state using a stable isotopically labelled microtracer approach.

Participants will take alectinib-d6 (microtracer) with and without food on different days.

DETAILED DESCRIPTION:
The aim of this study is to determine the food-effect of a standardized Dutch breakfast on the pharmacokinetics of alectinib. Despite the fact that three studies have reported a food-effect on alectinib pharmacokinetics, it is still unclear what the food-effect is on alectinib exposure in the daily lives of patients. It is important to understand this effect due the high inter- and intra-individual variability observed in alectinib exposure as well as the observed exposure-response relationship. Food might be a strategy to increase exposure without dose increase or reduce intra-individual variability.

A conventional, cross-over, food-effect study requires the participating patients to administer the investigational drug with and without food over several days until steady-state is reached (approximately 5 times the half-life of the respective drug). When steady-state is reached, blood samples will be collected for the determination of exposure of the investigational drug. However, this study design is inappropriate for the determination of the food-effect of alectinib due to possibly underexposure. A previously reported exposure-response analysis reported significantly decreased survival for NSCLC patients with an alectinib trough plasma concentrations (Ctrough) <435 ng/mL. Clinical trial simulations demonstrated that 55.5% of patients will have Ctrough below the target when alectinib is administered under fasting conditions assuming a food-effect of 40%.

A microtracer approach was chosen to determine the food-effect on alectinib pharmacokinetics without influencing the therapeutic treatment. A microtracer is a 100 µg dose of a stable isotopically labelled (SIL) drug. These microtracers have been used for the determination of absolute food-effect. Due to the mass difference between the therapeutic administered drug and the microtracer, the concentrations of both compounds can be simultaneously quantified in the same sample.

ELIGIBILITY:
Inclusion Criteria:

1. Currently treated with alectinib for NSCLC or other oncological indications;
2. On alectinib treatment at a stable dose of 600 mg twice daily (≥ 7 days) according to standard of care
3. Age ≥ 18 years;
4. Able and willing to give written informed consent;
5. world health organization (WHO) performance status of 0,1 or 2;
6. Able and willing to undergo blood sampling for pharmacokinetic analysis;
7. Able and willing to get one intravenous line for pharmacokinetic sampling
8. Able and willing to comply with study restrictions and to remain at the study center for the required duration.
9. Able and willing to undergo the defined food interventions

Exclusion Criteria:

1. Any treatment with investigational drugs (alectinib-d6) within 30 days or 5 half-lives prior to receiving the investigational treatment;
2. Any treatment with inhibitors of CYP3A4 (e.g. boceprevir, clarithromycin, erythromycin, indinavir, itraconazole, ketoconazole, ritonavir and voriconazole), inhibitors of Pgp (e.g. cyclosporine, kinidine, and verapamil), inhibitors of breast cancer resistance protein (BCRP) (e.g. lapatinib), inductors of CYP3A4, Pgp or BCRP;
3. Patients suffering from any known disease or dysfunction that might influence the dissolution and/or absorption of alectinib (e.g. inflammatory bowel disease, gastric bypass).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
food-effect on alectinib | 10 days
  To determine the food-effect of a standardised Dutch breakfast on the pharmacokinetics (Cmax) of oral alectinib (Alecensa®), at steady state using a stable isotopically labelled microtracer approach.
food-effect on alectinib | 10 days
  To determine the food-effect of a standardised Dutch breakfast on the pharmacokinetics (AUC and relative bioavailability (F)) of oral alectinib (Alecensa®), at steady state using a stable isotopically labelled microtracer approach.
  looking at Cmax

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands